CLINICAL TRIAL: NCT06968000
Title: Pilot, Controlled, Double-blind Study to Evaluate the Effect of the Exposome Anionic Enrichment System (Biow) on Hospital Recovery Quality, Clinical Response, and Sleep Quality in Postoperative Patients
Brief Title: Double-blind Pilot Study on the Effect of Anionic Exposome Enrichment (Biow) on Recovery and Sleep Quality in Postoperative Patients
Acronym: EOX
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: EOX - BIOW
Record Dates: First submitted 2025-05-05; First posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2024-10

CONDITIONS: Inflammatory Response After Surgery; Postoperative Recovery
Keywords: Exposome; Bioavailable anions; Postoperative recovery; Mitochondrial function; Oxidative stress; Surgical inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a quadruple-blind study (participant, care provider, investigator, outcomes assessor). The masking is ensured by installing EOX devices in all rooms, regardless of group allocation. Devices appear identical, emit no distinguishable noise, light, or heat, and all display a powered-on light indicator. Only the manufacturer knows which units are active or inactive (placebo). Room assignment is determined by hospital admission scheduling, not influenced by study personnel. Neither patients nor clinical or research staff are aware of the device's operational status, ensuring complete masking throughout the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active mode (Active Comparator): Device: EOX (active mode)
  Dose/Duration: 96 hours of continuous exposure in the hospital room
  Frequency: Continuous (24h/day during hospitalization)
  Interventions: Device: EOX Anion-Enriched Hospital Room
- Inactive mode (Sham Comparator): Intervention:
  Device: EOX (inactive mode)
  Dose/Duration: 96 hours in the hospital room
  Frequency: Device is present but non-functional (placebo exposure)
  Interventions: Device: EOX Anion-Enriched Hospital Room

INTERVENTIONS:
Device: EOX Anion-Enriched Hospital Room — Participants are assigned to hospital rooms equipped with an operational EOX device, which actively regenerates air and releases bioavailable anions through cold atmospheric plasma. Exposure lasts for 96 hours postoperatively. The intervention aims to enhance postoperative recovery by modulating oxidative stress, improving mitochondrial function, and promoting sleep quality.

SUMMARY:
Airborne nanoparticle exposure is increasingly recognized as a significant contributor to oxidative stress, mitochondrial dysfunction, and low-grade systemic inflammation-factors that impair postoperative recovery. The World Health Organization and European initiatives such as the Human Exposome Project have highlighted the clinical importance of the exposome, defined as the totality of environmental exposures influencing health throughout life.

EOX is a CE-certified air regeneration system designed to modify the indoor exposome through a dual mechanism: advanced filtration and controlled emission of bioavailable anions using cold atmospheric plasma (CAP). Its multistage filter removes particulate matter, pathogens, and volatile organic compounds, while the anionic plasma phase modulates cellular oxidative balance and metabolic function.

Experimental and clinical data indicate that exposure to EOX improves mitochondrial efficiency, increases ATP production, and reduces oxidative protein damage. EOX has also been shown to influence molecular pathways involved in stress adaptation and repair, such as the HIF-1α-VEGF-EPO axis and protein synthesis signaling (e.g., mTOR-p70S6K). These mechanisms may collectively enhance tissue recovery, vascularization, and metabolic resilience in the postoperative setting.

The present study investigates the effects of EOX in hospitalized postoperative patients, evaluating both subjective (sleep quality, well-being) and objective (vital signs, metabolomics, microbiota composition) endpoints. The central hypothesis is that EOX induces a beneficial hormetic response-an adaptive reaction to mild environmental stressors-reflected by improved clinical recovery and biomarker modulation (e.g., succinate reduction, increased ATPase activity). The goal is to assess whether EOX can serve as an effective environmental intervention to support physiological healing and improve the quality of inpatient recovery.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥18 years, regardless of sex.
* Undergoing elective general surgery, preferably hepatobiliary procedures.
* Hospitalized for at least 4 days postoperatively in Unit 69 (HUFJD).
* Able to provide written informed consent.
* Considered to have medium or high risk of oxidative stress or mitochondrial dysfunction.

Exclusion Criteria:

* Surgery within the previous 6 months, either outpatient or inpatient.
* Diagnosed psychiatric or neurological disorders, including epilepsy.
* Active progressive cancer or chronic inflammatory disease.
* Cognitive impairment or inability to comply with study procedures.
* BMI ≥30 kg/m² (obesity class I or higher).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Hormetic clinical response associated with EOX exposure during the first 96 hours post-surgery | Baseline (day 0) to 96 hours post-intervention
  Evaluation of the adaptive (hormetic) biological response induced by anion-enriched air using EOX. This will be assessed through:
  * 10% increase in plasma ATPase activity, and/or
  * 10% decrease in plasma succinate levels, and/or
  * 10% increase in uninterrupted sleep hours (based on sleep diary and nursing records), during the 96-hour postoperative hospital stay.

CONTACTS AND LOCATIONS:
Locations (1):
- Fundacion Instituto de Investigacion Sanitaria Fjd, Madrid, Madrid, Spain

REFERENCES:
- [Background] Cortazar OD, Megia-Macias A, Moreno S, Brun A, Gomez-Casado E. Vulnerability of SARS-CoV-2 and PR8 H1N1 virus to cold atmospheric plasma activated media. Sci Rep. 2022 Jan 7;12(1):263. doi: 10.1038/s41598-021-04360-y. PMID 34997166
- [Background] Antuna E, Carlos Bermejo-Millo J, Caso-Onzain E, Caso-Pelaez E, Potes Y, Coto-Montes A. Removal of Environmental Nanoparticles Increases Protein Synthesis and Energy Production in Healthy Humans. Front Bioeng Biotechnol. 2022 Feb 14;10:800011. doi: 10.3389/fbioe.2022.800011. eCollection 2022. PMID 35237574